CLINICAL TRIAL: NCT00568048
Title: Temozolomide Combined With Bevacizumab in Metastatic Melanoma. A Multicenter Phase II Trial
Brief Title: Temozolomide and Bevacizumab in Treating Patients With Stage IV Melanoma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 50/07; SWS-SAKK-50/07; EU-20790; CDR0000577499
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Bevacizumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination Therapy Temozolomide & Bevacizumab (Experimental): Combination therapy
  * Temozolomide 150 mg/m2 p.o., days 1-7, repeated every 14 days
  * Bevacizumab 10 mg/kg i.v., day 1, repeated every 14 days
  Interventions: Biological: bevacizumab; Drug: temozolomide

INTERVENTIONS:
Biological: bevacizumab — 10 mg/kg i.v., on day 1 of every cycle (14 days) until PD or any other event qualifying for stopping treatment
  Other Names: Avastin
Drug: temozolomide — 150 mg/m2 p.o., on days 1-7 of every cycle (14 days) until PD or any other event qualifying for stopping treatment
  Other Names: Temodal

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving temozolomide together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving temozolomide together with bevacizumab works in treating patients with stage IV melanoma that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy of temozolomide in combination with bevacizumab in patients with unresectable stage IV melanoma.

Secondary

* To evaluate the safety and tolerability of this regimen.

Tertiary

* To evaluate the prognostic and predictive significance of circulating endothelial cells and endothelial progenitor cells in patients treated with this regimen.
* To predict tumor response and outcome in patients treated with this regimen by measuring hypermethylation of the tumor.

OUTLINE: This is a multicenter study.

Patients receive oral temozolomide once daily on days 1-7 and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

Blood is collected at baseline and on day 1 of course 2. Samples are analyzed for circulating endothelial cells and endothelial progenitor cells by flow cytometry and pro- and anti-angiogenic serum factors by ELISA. Paraffin-embedded tumor tissue is analyzed for MGMT promoter methylation status by methylation-specific PCR; MGMT protein expression by IHC; and MSH2, MSH6, and MLH-1 expression (DNA repair enzymes).

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma

  * Unresectable stage IV disease
  * Mucosal and unknown primary disease allowed
* Measurable disease, defined as at least one lesion that can be measured in at least one dimension as ≥ 20 mm (or as ≥ 10 mm if the CT slice thickness is ≤ 5 mm)

  * Measurable lesion must be outside a previously treated area
* Must have 1 paraffin block of primary tumor and/or metastatic tissue available for analysis of MGMT
* No ocular melanoma
* No bleeding skin metastases
* No CNS metastases (even if previously treated) by brain MRI

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* ANC ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Hemoglobin ≥ 90 g/L (transfusion allowed)
* Serum total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and alkaline phosphatase ≤ 2.5 times ULN (5 times ULN in patients with liver metastases)
* Serum creatinine < 177 μmol/L
* Proteinuria < 2+ by urine dipstick OR urine protein ≤ 1 g by 24-hour urine collection
* INR ≤ 1.5
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study treatment
* No other primary tumors within the past 5 years, except adequately controlled limited basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No history or evidence of CNS disease unrelated to cancer (e.g., uncontrolled seizures) by physical/neurological examination, unless adequately treated with standard medical therapy
* No frequent vomiting or any other pre-existing medical condition that would preclude swallowing and/or absorption of oral medication
* No history or evidence of inherited bleeding diathesis or coagulopathy with risk of bleeding
* No uncontrolled hypertension (i.e., systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 100 mm Hg, measured repeatedly, despite adequate treatment with at least two different antihypertensive drugs)
* No clinically significant (i.e., active) cardiovascular disease, including any of the following:

  * Cerebrovascular accident/stroke or myocardial infarction within the past 6 months
  * Unstable angina
  * New York Heart Association (NYHA) class II or greater congestive heart failure
  * Serious cardiac arrhythmia (i.e., ventricular arrhythmia, high-grade atrioventricular-block) that requires medication during the study, interferes with regularity of the study treatment, or is uncontrolled by medication
* No serious non-healing wound, active peptic ulcer, or non-healing bone fracture
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No significant traumatic injury within the past 30 days
* No uncontrolled active infection
* No known HIV infection
* No known hypersensitivity to any of the study drugs or excipients
* No evidence of any other disease, metabolic or psychological dysfunction, psychiatric disorder, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, or that may affect patient compliance with study routines, or places the patient at high risk from treatment-related complications

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior adjuvant cytokine therapy (e.g., interleukin, interferon) or vaccine therapy and recovered

  * Prior vaccine therapy for stage IV disease allowed
* Prior perfusion therapy (limb and liver) for loco-regional disease allowed
* No prior chemotherapy for metastatic disease
* No prior bevacizumab or other angiogenic inhibitors
* No prior radiotherapy to lesion(s) selected for measurement
* More than 30 days since prior treatment in a clinical trial
* More than 30 days since prior major surgery with high risk of bleeding
* More than 24 hours since prior minor surgery
* More than 10 days since prior and no concurrent full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes

  * Prophylactic use of anticoagulants is allowed (e.g., maintenance of venous catheter)
* More than 10 days since prior and no concurrent acetylsalicylic acid (> 325 mg/day) or clopidogrel (> 75 mg/day)
* No other concurrent non-steroidal anti-inflammatory drugs (NSAIDs)
* No concurrent dipyridamole
* No concurrent major surgery
* No concurrent radiotherapy to the target lesions
* No other concurrent experimental drugs or anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-12; Primary Completion 2010-12 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Clinical benefit number of patients with complete response [CR], partial response [PR], or stable disease) according to RECIST criteria | at 12 weeks

SECONDARY OUTCOMES:
Best overall response (CR, PR) according to RECIST criteria | from trial treatment start until PD
Duration of response | time from disease stabilisation until PD
Progression free survival | time from trial registration until disease progression or death
Overall survival | time from trial registration until death
Adverse events | time from start trial treatment until 30 days after treatment stop. Adverse events will be assessed according to NCI CTCAE v3.0.

CONTACTS AND LOCATIONS:
Overall Officials: Roger von Moos, MD, Study Chair — Kantonsspital Graubuenden
Locations (1):
- Kantonsspital Graubuenden, Chur, Switzerland

REFERENCES:
- [Result] von Moos R, Seifert B, Simcock M, Goldinger SM, Gillessen S, Ochsenbein A, Michielin O, Cathomas R, Schlappi M, Moch H, Schraml PH, Mjhic-Probst D, Mamot C, Schonewolf N, Dummer R; Swiss Group for Clinical Cancer Research (SAKK). First-line temozolomide combined with bevacizumab in metastatic melanoma: a multicentre phase II trial (SAKK 50/07). Ann Oncol. 2012 Feb;23(2):531-6. doi: 10.1093/annonc/mdr126. Epub 2011 Apr 28. PMID 21527587
- [Result] Dummer R, Michielin O, Seifert B, et al.: First-line temozolomide (TEM) combined with bevacizumab (BEV) in metastatic melanoma (MM): A multicenter phase II trial (SAKK 50/07). [Abstract] J Clin Oncol 28 (Suppl 15): A-8521, 2010.
- [Result] Fuerstenberger G, Boneberg E, Simcock M, et al.: Predictive and prognostic potential of angiogenic serum factors and circulating endothelial cells in metastatic melanoma patients receiving temozolamide plus bevacizumab (SAKK 50/07). [Abstract] J Clin Oncol 28 (Suppl 15): A-8585, 2010.
- [Result] Schraml P, von Teichman A, Mihic-Probst D, Simcock M, Ochsenbein A, Dummer R, Michielin O, Seifert B, Schlappi M, Moch H, von Moos R. Predictive value of the MGMT promoter methylation status in metastatic melanoma patients receiving first-line temozolomide plus bevacizumab in the trial SAKK 50/07. Oncol Rep. 2012 Aug;28(2):654-8. doi: 10.3892/or.2012.1826. Epub 2012 May 18. PMID 22614944